CLINICAL TRIAL: NCT00134160
Title: The Study Comparing the Incidence of Cardiovascular Events Between High-dose ARB Monotherapy and Combination Therapy With ARB and Calcium Channel Blocker in Japanese Elderly Hypertensive Patients at High Cardiovascular Risk
Brief Title: OlmeSartan and Calcium Antagonists Randomized (OSCAR) Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OSCAR Study (Other)
Collaborators: Japan Heart Foundation (Other)
Responsible Party: Ogawa Hisao, Kumamoto University Graduate School of Medical Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15-April-2005
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: Aged; Hypertension; Cardiovascular Diseases; Angiotensin II Type 1 Receptor Blockers; Calcium Channel Blockers; Combination Drug Therapy; Diabetes Mellitus Type 2
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Diabetes Mellitus, Type 2 | interventions — Olmesartan Medoxomil; Calcium Channel Blockers; Amlodipine; azelnidipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): High-dose ARB monotherapy
  Interventions: Drug: Olmesartan medoxomil
- 2 (Active Comparator): Combination therapy of ARB with Calcium Channel Blocker
  Interventions: Drug: Calcium channel blockers (amlodipine, azelnidipine)

INTERVENTIONS:
Drug: Olmesartan medoxomil — Olmesartan medoxomil 40mg/Day
  Arms: 1
Drug: Calcium channel blockers (amlodipine, azelnidipine) — Olmesartan medoxomil 20mg/Day with Calcium channel blockers (amlodipine or azelnidipine)
  Arms: 2

SUMMARY:
The purpose of this study is to investigate whether high-dose angiotensin II receptor blocker (ARB) monotherapy or combination therapy with ARB and calcium channel blockers is more effective in reducing the incidence of cardiovascular events in Japanese elderly high-risk hypertensive patients not adequately controlled by standard dose ARB alone.

DETAILED DESCRIPTION:
Hypertension is one of the major risk factors of cardiovascular diseases. It is also important for elderly hypertensive patients to strictly reduce their blood pressures to prevent cardiovascular events. Although angiotensin II receptor blockers (ARBs) are increasingly used in antihypertensive treatment recently, few studies have been performed in Japan to assess the difference between high-dose ARB monotherapy and combination therapy of ARB with calcium channel blocker (CCB) in prevention of cardiovascular diseases for patients whose blood pressure is not well controlled by ARB monotherapy. OSCAR-study is a multicenter, active-controlled, 2-arm parallel group comparison, prospective randomized open blinded end-point (PROBE) design study. The dose administered is olmesartan medoxomil 20mg/day as ARB monotherapy in the 'Step 1' period. If the blood pressure is not adequately controlled and treatment is well tolerated then the dose is changed to olmesartan medoxomil 40mg/day in the high-dose ARB monotherapy group, or olmesartan medoxomil 20mg/day and a CCB in the combination therapy group in the 'Step 2' period. At least 500 patients will be enrolled in each group, and the follow-up duration will be 3 years. The primary objective is to compare the incidence of a composite of fatal and non-fatal cardiovascular events, and all cause mortality between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 65 years or older, and less than 85 years (at the time of informed consent), regardless of sex
* Current antihypertensive treatment with monotherapy
* SBP ≥ 140mmHg or DBP ≥ 90mmHg in a sitting position on two measurements on two clinic visits
* At least one of the following risk factors:

  * Diabetes mellitus Type 2;
  * History of cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage, or transient ischemic attack (more than 6 months before giving informed consent);
  * Diagnosis of asymptomatic cerebrovascular disease;
  * History of myocardial infarction (more than 6 months before giving informed consent);
  * Diagnosis of angina pectoris or heart failure (New York Heart Association [NYHA] functional classification I or II);
  * Diagnosis of left ventricular hypertrophy (thickness of the wall of interventricular septum ≥ 12mm on echocardiography or Sv1+Rv5 ≥ 35mm on electrocardiography before informed consent);
  * Diagnosis of aortic aneurysm;
  * History of aortic dissection (more than 6 months before giving informed consent);
  * Diagnosis of arteriosclerotic peripheral arterial obstruction (Fontaine classification from 2 to 4);
  * Serum creatinine: 1.2-2.5mg/dL (male); 1.0-2.5mg/dL (female);
  * Proteinuria: ≥ +1 (or ≥ 0.3g/g･Cr. estimated from 24-hour urine collection or random urinary protein corrected by urine creatinine).

Exclusion Criteria:

* Secondary hypertension or malignant hypertension
* Heart failure (NYHA functional classification III or IV)
* Required treatment for malignant tumor
* Serious liver or renal dysfunction (serum creatinine > 2.5mg/dL or with dialysis treatment)
* Not appropriate for change to the test drugs from current therapy for hypertension or coronary diseases (i.e. calcium channel blockers, β-blockers, thiazide diuretics, etc.)
* History of serious adverse drug reactions to angiotensin II receptor blockers or calcium channel blockers
* Patients with other serious reasons (i.e. illness, significant abnormalities, etc.) that investigators judge inappropriate for the study

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2005-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
A composite of fatal and non-fatal cardiovascular events: Cerebrovascular events (cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage, stroke of undetermined etiology and transient ischemic attack) | 36 Months
Coronary events (sudden death, myocardial infarction, angina pectoris, asymptomatic myocardial ischemia) | 36 Months
Heart failure | 36 Months
Vascular events (aortic aneurysm, aortic dissection, and arteriosclerotic diseases) | 36 Months
Diabetic complications (nephropathy, retinopathy and neuropathy) | 36 Months
Renal dysfunction (doubling of serum creatinine, end stage renal diseases) | 36 Months
All cause mortality | 36 Months

SECONDARY OUTCOMES:
Development of each cardiovascular event | 36 Months
Blood pressure change (systolic blood pressure [SBP], diastolic blood pressure [DBP], mean blood pressure [MBP]) at every observation point in the follow-up period | 36 Months
Serious adverse events other than primary outcome events | 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Kikuo Arakawa, MD, Study Chair — Emeritus Professor Fukuoka University, Fukuoka, Japan
Locations (2):
- Japan (2):
  - Department of Cardiovascular Medicine Graduate School of Medical Science Kumamoto University, 1-1-1 Honjyo, Kumamoto-City, Kumamoto
  - OSCAR-Study Data Center, ShinjukuParkTower30FN, 3-7-1 Nishi-Shinjuku, Shinjuku-ku, Tokyo

REFERENCES:
- [Derived] Do DV, Han G, Abariga SA, Sleilati G, Vedula SS, Hawkins BS. Blood pressure control for diabetic retinopathy. Cochrane Database Syst Rev. 2023 Mar 28;3(3):CD006127. doi: 10.1002/14651858.CD006127.pub3. PMID 36975019
- [Derived] Kim-Mitsuyama S, Ogawa H, Matsui K, Jinnouchi T, Jinnouchi H, Arakawa K; OSCAR Study Group. Differential effectiveness of ARB plus CCB therapy and high-dose ARB therapy in high-risk elderly hypertensive patients: subanalysis of the OSCAR study. Hypertens Res. 2015 Mar;38(3):199-207. doi: 10.1038/hr.2014.164. Epub 2014 Dec 4. PMID 25471234
- [Derived] Matsui K, Kim-Mitsuyama S, Ogawa H, Jinnouchi T, Jinnouchi H, Arakawa K; OlmeSartan Calcium Antagonists Randomized (OSCAR) Study Group. Sex differences in response to angiotensin II receptor blocker-based therapy in elderly, high-risk, hypertensive Japanese patients: a subanalysis of the OSCAR study. Hypertens Res. 2014 Jun;37(6):526-32. doi: 10.1038/hr.2014.23. Epub 2014 Mar 6. PMID 24599010
- [Derived] Kim-Mitsuyama S, Ogawa H, Matsui K, Jinnouchi T, Jinnouchi H, Arakawa K. An angiotensin II receptor blocker-calcium channel blocker combination prevents cardiovascular events in elderly high-risk hypertensive patients with chronic kidney disease better than high-dose angiotensin II receptor blockade alone. Kidney Int. 2013 Jan;83(1):167-76. doi: 10.1038/ki.2012.326. Epub 2012 Oct 10. PMID 23051740
- [Derived] Ogawa H, Kim-Mitsuyama S, Matsui K, Jinnouchi T, Jinnouchi H, Arakawa K; OlmeSartan and Calcium Antagonists Randomized (OSCAR) Study Group. Angiotensin II receptor blocker-based therapy in Japanese elderly, high-risk, hypertensive patients. Am J Med. 2012 Oct;125(10):981-90. doi: 10.1016/j.amjmed.2011.12.010. Epub 2012 Apr 14. PMID 22503610
- [Derived] Ogawa H, Kim-Mitsuyama S, Jinnouchi T, Matsui K, Arakawa K. Rationale, design and patient baseline characteristics of OlmeSartan and calcium antagonists randomized (OSCAR) study: a study comparing the incidence of cardiovascular events between high-dose angiotensin II receptor blocker (ARB) monotherapy and combination therapy of ARB with calcium channel blocker in Japanese elderly high-risk hypertensive patients (ClinicalTrials. gov no. NCT00134160). Hypertens Res. 2009 Jul;32(7):575-80. doi: 10.1038/hr.2009.60. Epub 2009 May 15. PMID 19444280